CLINICAL TRIAL: NCT01911533
Title: Veno-venous Extracorporeal CO2 Removal in ARDS-patients to Treat Respiratory Acidosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/505
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: ACUTE RESPIRATORY DISTRESS SYNDROME
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- extracorporeal CO2 (Experimental)
  Interventions: Procedure: extracorporeal removal of CO2 (ECCO2-R); Procedure: No extracorporeal CO2-removal

INTERVENTIONS:
Procedure: extracorporeal removal of CO2 (ECCO2-R) — To promote a better gas-exchange, the patient with ARDS will be mechanically ventilated. This can be aggressive and harmful for the lungs. With the use of an extra-corporeal CO2-remover, CO2 can be removed so that the mechanical ventilation setting will be less aggressive and will decrease lesions in the lung. The veno-venous extracorporeal CO2-remover pumps blood from a vein via a catheter through an oxygenator (gas exchanger that adds oxygen to the blood and extracts carbon dioxide from the blood) and back into a vein.
Procedure: No extracorporeal CO2-removal — Patients are their own control group.

SUMMARY:
Hypothesis:

Extracorporeal removal of CO2 can treat hypercapnia and respiratory acidosis, which allows application of lung protective ventilation. This downgrading of mechanical ventilation promotes better and more quickly lung recovery.

Aim:

The aim of the study is to treat respiratory acidosis and to reduce plateau pressures by using an extracorporeal removal of CO2 (ECCO2-R).

This prospective study will include 10 patients with an Acute Respiratory Distress Syndrome (ARDS). ARDS is an inflammatory response in the lungs, the onset is acute with pulmonary oedema and shows bilateral densities on chest radiography. The take up of oxygen and the loss of CO2 in the lungs are difficult. Moreover the patient's blood can become acidic due to too much CO2.

To promote a better gas-exchange, the patient with ARDS will be mechanically ventilated. This can be aggressive and harmful for the lungs. With the use of an extra-corporeal CO2-remover, CO2 can be removed so that the mechanical ventilation setting will be less aggressive and will decrease lesions in the lung. The veno-venous extracorporeal CO2-remover pumps blood from a vein via a catheter through an oxygenator (gas exchanger that adds oxygen to the blood and extracts carbon dioxide from the blood) and back into a vein.

The investigators will use a standard dialysis catheter that will be put in a large vein. To prevent clotting of the system, the patient will receive heparin.

In the study the investigators will work in periods of two hours, the situation before and after carbon dioxide removal will be compared. With this study the investigators want to prove that the CO2 in the blood decreases with at least 20 % with the use of the extracorporeal CO2 remover. More over the investigators want to prove that lower mechanical ventilation settings (thanks to CO2-removal by the ECCO2-R) will produce fewer lesions to the lungs.

ELIGIBILITY:
Inclusion criteria:

* Acute onset of ARDS criteria on chest X-ray or CT scan
* Moderate (PaO2/ FiO2 <200) or severe ARDS (PaO2/ FiO2 <100) (FiO2: fraction of inspired oxygen)
* Respiratory acidosis with pH< 7,25,
* With plateau pressure of 28cmH20 or higher,

Exclusion criteria:

* <18 years of age
* Pregnancy
* Obesity with BMI> 30
* Contraindication for anticlotting therapy
* Chest wall abnormalities
* No presumed consent of representatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2014-06-12 (Actual); Study Completion 2014-09-12 (Actual)

PRIMARY OUTCOMES:
To obtain a reduction of 20% in arterial partial CO2 pressure (PaCO2) after the first two hours of ECCO2-R therapy. | After the first two hours of ECCO2-R therapy, every 2 hours for a maximum of 5 days.
  Arterial blood gasses, ventilator settings will be measured.

SECONDARY OUTCOMES:
Reduction in Plateau pressures to levels between 25 and 28 cm H2O. | Every 2 hours during procedure for a maximum of 5 days.
  Arterial blood gasses and ventilator settings will be measured.
• Reduction in tidal volumes to 6ml/kg predicted body weight (PBW) or lower, with a minimum of 3ml/kg PBW. | Every 2 hours during the procedure for a maximum of 5 days.
  Arterial blood gasses and ventilator settings will be measured.
Increase in pH to the normal range of 7,35 to 7,45. | Every 2 hours during the procedure for a maximum of 5 days.
  Arterial blood gasses and ventilator settings will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Harlinde Peperstraete, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Peperstraete H, Eloot S, Depuydt P, De Somer F, Roosens C, Hoste E. Low flow extracorporeal CO2 removal in ARDS patients: a prospective short-term crossover pilot study. BMC Anesthesiol. 2017 Nov 28;17(1):155. doi: 10.1186/s12871-017-0445-9. PMID 29179681
- See also: Related Info — http://www.uzgent.be